CLINICAL TRIAL: NCT02851004
Title: A Phase Ib/II Study of BBI608 in Combination With Pembrolizumab in Patients With Metastatic Colorectal Cancer
Brief Title: Special Combination of BBI608 and Pembrolizumab
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: On the request of the investigational drug provider. No subjects were newly enrolled in the additional cohort as they were preparing to resume enrollment in the additional cohort. Currently, it is preparing the creation of clinical study report.
Sponsor: Takayuki Yoshino (Other)
Collaborators: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Takayuki Yoshino, Director of Gastrointestinal Oncology Division, National Cancer Center Hospital East
Organization: National Cancer Center Hospital East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC1503
Record Dates: First submitted 2016-07-14; First posted 2016-08-01 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — napabucasin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: [Phase Ib] 6 to 9 patients
  [Phase II] Cohort A (MSI-H): 10 patients Cohort B (MSS): 40 patients Including patients with metastatic CRC treated at the recommended dose (RD) level in the Phase Ib part who meet criteria for the full analysis set (FAS)
  [Additional cohort to the Phase II part]
  1. st stage: CMS 1 or 4, MSS right-side colon cancers*: 10 patients
  2. nd stage:
     1. : If no patient shows a partial or complete response in the 1st stage, the study will be prematurely terminated.
     2. : If 1 or 2 patients show a partial or complete response in the 1st stage, 19 patients with CMS 1 or 4, MSS right-side colon cancers will be enrolled additionally.
     3. : If 3 or more patients show a partial or complete response in the 1st stage, 19 patients with CMS 1 or 4, MSS right-side colon cancers and 10 patients with CMS 1 or 4, MSS left-side colon cancers* will be enrolled additionally.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BBI608 + Pembrolizumab (Experimental): BBI608 and Pembrolizumab
  Interventions: Drug: Napabucasin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Napabucasin — 1 cycle is 21days.
  BBI608: Oral administration at a dose of 240mg or 480 mg twice daily (BID), every day.
  [Additional cohort to the Phase II part] Oral administration at a dose of 240mg mg BID, every day
  The therapy will be repeated until meeting the discontinuation criteria.
Drug: Pembrolizumab — 1 cycle is 21days.
  Pembrolizumab: Administration at a dose of 200 mg/body on Day 1 of each cycle
  [Additional cohort to the Phase II part] Administration at a dose of 200 mg/body on Day 1 of each cycle.
  The therapy will be repeated until meeting the discontinuation criteria.

SUMMARY:
the efficacy and safety of BBI608 in combination with pembrolizumab

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase Ib/II study to exploratively evaluate the efficacy and safety of BBI608 in combination with pembrolizumab in patients with metastatic colorectal cancer (CRC) not responded to or intolerant of standard chemotherapy.The same analysis will be performed for the additional cohort to the Phase II part, consisting of patients with metastatic CMS 1 or 4, MMS, CRC not responsive to or intolerant of standard chemotherapy.

ELIGIBILITY:
For the additional cohort to the Phase II part, screening tests will be performed to identify CMS 1 or 4 and MSS before obtaining informed consent.

Patients, who meet all of the following inclusion criteria and none of the exclusion criteria, are eligible for enrollment in the study.

Inclusion Criteria

1. Patients who personally provided written consent to be the subjects of the study
2. Age of 20 years or older on the day of informed consent
3. [Phase Ib] Histologically confirmed gastrointestinal cancer

   [Phase II] Histologically confirmed colon or rectal cancer that is adenocarcinoma , and identification of at least the KRAS codon 12 and 13 mutation status determined by RAS gene testing. Confirmation of the microsatellite instability (MSI) status.

   [Additional cohort to the Phase II part] Histologically confirmed colon or rectal cancer that is adenocarcinoma, and identification of RAS mutation status. Identification of CMS 1 or 4 and MSS by screening tests.
4. [Phase Ib] Gastrointestinal cancer not responded to or intolerant of standard chemotherapy

   [Phase II]A history of treatment with one or more regimens of the following standard chemotherapies for metastatic CRC, and being not responded to or tolerated the chemotherapies

   [Additional cohort to the Phase II part] In accordance with Cohort B in the Phase II part.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1
6. Patients with evaluable lesions (Cohort A in Phase II and Phase Ib) or measurable lesions (Cohort B in Phase II and the additional cohort to the Phase II part) specified in the RECIST version 1.1
7. Patients with adequate organ function based on the following laboratory values measured within 7 days before enrollment
8. Women of childbearing potential who are negative in a pregnancy test within 7 days before enrollment. Both male and female patients who consent to practice appropriate contraception during the study and for 4 months after the discontinuation of the protocol treatment
9. Patients with an expected survival of at least 3 months

Exclusion criteria

1. Patients who received chemotherapy, molecular-targeted agents and/or palliative radiotherapy within 2 weeks before the start of the protocol treatment or have not recovered from toxicity caused by previous treatment
2. Patients who underwent general anesthesia, surgery requiring hospitalization and extensive radiotherapy within 4 weeks before the start of the protocol treatment or minor surgery such as implantation of a central venous access device within two weeks before the start of the protocol treatment
3. Patients with active central nervous system metastases or carcinomatous meningitis.
4. Pregnant or lactating women
5. Patients who are unable or not willing to take BBI608 capsules every day
6. Patients with gastrointestinal disease markedly interfering with the absorption of oral formulations as judged by the investigator
7. Patients with active autoimmune disease requiring systemic treatment within 2 years before the start of the protocol treatment.
8. Patients with a history or signs of interstitial lung disease or active non-infectious pneumonitis
9. Patients who underwent organ or bone marrow transplantation
10. Patients who received a live vaccine within 30 days before the start of the protocol treatment
11. Patients who participated in another clinical study within 4 weeks before the start of the protocol treatment and used or using an investigational drug or device
12. Patients who previously received immunotherapy with drugs targeting PD-1, PD-L1 and/or PD-L2 or BBI608 therapy, or took part in a clinical study of pembrolizumab or BBI608
13. Patients with uncontrollable complications
14. Patients with a history of other malignancies within 3 years before the start of the protocol treatment.
15. Patients with clinically significant Electrocardiogram (ECG) abnormalities
16. Patients with a history of Human Immunodeficiency Virus (HIV)
17. Patients with active hepatitis B or C

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
irORR | 2 years
  Immune-related objective response rate determined by their Response Evaluation Criteria In Solid Tumors (RESIST): for the Phase II part
ORR | 1 year
  Objective response rate determined by RECIST version 1.1: for additional cohort to the Phase II part

SECONDARY OUTCOMES:
irPFS | 12 weeks
  Immune-related progression free survival rate at week 12 determined by the irRECIST
ORR | 2 years
  Objective response rate determined by RECIST version 1.1: for the Phase II part
irORR | 1 year
  Immune-related objective response rate determined by their Response Evaluation Criteria In Solid Tumors (RESIST): for additional cohort to the Phase II part
Progression free survival rate at week 12 determined by the RECIST version 1.1 | 12 weeks
  PFS
PFS | 3 years
  Progression free survival
OS | 4 years
  Overall survival
DCR | 2 years
  Disease Control rate
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 4 years
  Incidence of adverse events
Pharmacokinetic | 2 months
  Area under the blood concentration-time curve (AUC)
Pharmacokinetic | 2 months
  CmaxPeak Plasma Concentration (Cmax)

OTHER OUTCOMES:
efficacy according to immune status - Immune status will be analyzed using biopsy and blood samples by flow cytometry, RNA seq, whole exome sequencing, and immunohistochemistry etc. | 3 years
  Efficacy evaluations according to immune status
safety according to immune status | 3 years
  Safety evaluations according to immune status

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Yoshino, Dr, Study Chair — National Cancer Center Hospital East
Locations (1):
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No